CLINICAL TRIAL: NCT02790268
Title: Ultrasound Biomicroscopic Analysis of Cionni Ring and In-the-bag IOL Implantation for Subluxated Lenses
Status: Completed | Type: Observational
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, Director, Iladevi Cataract and IOL Research Center, Iladevi Cataract and IOL Research Center
Other Study IDs: ICIRC-UBM
Record Dates: First submitted 2016-05-24; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Lens Subluxation
Keywords: Cionni Ring; Ultrasound Biomicroscopy
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lens Subluxation: Pediatric eyes with lens subluxation undergoing Cionni Ring Bag fixation with in-the-bag IOL Implantation
  Interventions: Procedure: Lens Subluxation Surgery

INTERVENTIONS:
Procedure: Lens Subluxation Surgery — Surgical Intervention to include Cionni Ring implantation and in-the-bag IOL implantation

SUMMARY:
To report the Ultrasound Biomicroscopic findings following Cionni Ring bag fixation and in-the-bag IOL Implantation. To assess the relationship of the Bag and Cionni ring positioning in relation to surrounding ocular structures, in pediatric eyes

DETAILED DESCRIPTION:
Cionni ring fixation of the capsular bag in conjunction with placement of an IOL has been found to be safe and effective compared with other current alternatives, even given the exceptionally high difficulty levels and complexity of these cases, in both adult and pediatric eyes. One limitation of techniques requiring trans-scleral suturing is that the suture cannot always be passed under adequate visualization, and, once the knot is secured, the exact position of the Cionni ring cannot always be accurately localized. Analysis of Cionni ring position with respect to the IOL and iris is important, as faulty placement of the ring or IOL can lead to complications which can threaten vision, especially in children with a high predisposition towards postoperative adverse events. Unfortunately, pupillary dilatation and slit-lamp examination may not always be adequate to assess the Cionni ring or the eyelet position, as it occupies the peripheral section of the capsular bag. UBM has been shown to be accurate and reproducible in examining the haptic position in relation to the sulcus and ciliary body, anterior chamber depth (ACD), vitreous incarceration, focal iris abnormalities, angle anatomy, and relationship of the iris to the lens (straight or tilted). This study aims to provide information on UBM findings following Cionni ring implantation in pediatric eyes for non-traumatic subluxation of the crystalline lens.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years of age,
* Non-traumatic Lens Subluxation undergoing Cionni RIng Bag fixation with In-the-Bag IOL implantation

Exclusion Criteria:

* Traumatic Lens Subluxation
* Intraoperative inability to fixate the Cionni Ring

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing Cionni Ring Implantation with in-the-bag implantation for subluxated lenses
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ultrasound Biomicroscopic Measurement of Anterior Chamber Depth, Cionni Ring Position, distance from the posterior surface of iris and ciliary body region | 6 months postoperative
  To Measure in millimeters, the anterior chamber depth, the distance of cionni ring from posterior surface of iris, the distance of cionni ring from the ciliary body region

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Vasavada, MS,FRCS, Study Director — Iladevi Cataract & IOL Research Centre

IPD SHARING:
Plan to Share IPD: No